CLINICAL TRIAL: NCT03138642
Title: A Prospective Phase II Study in Patients With Mucosal Melanoma of Head and Neck in Intensity-modulated Radiotherapy Era
Brief Title: Mucosal Melanoma of Head and Neck in Intensity-modulated Radiotherapy Era
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lixia Lu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMHN-01
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Mucosal Melanoma
Keywords: mucosal melanoma; radiotherapy

STUDY DESIGN:
Intervention Model Description: All the patients receive extended resection to primary tumor and post-surgery RT. The patients are prescribed a EQD2 of 70-77Gy to GTV (residual tumor), 65-70Gy to CTV1(high-risk regions including tumor bed and gross macroscopic residual tumor), 50-55Gy to CTV2(low-risk regions) using Intensity-modulated radiotherapy (IMRT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RT (Experimental): The patients are prescribed a EQD2of 65-70Gy to CTV1(high-risk regions including tumor bed), 50-55Gy to CTV2(low-risk regions) using Intensity-modulated radiotherapy (IMRT). The Prophylactic irradiation to upper neck is is decided by radiation physicians and given a EQD2 of 70-77Gy to CTVnd (clinically negative lymph nodes), 50-55Gy to CTVn2（neck nodal regions). If there is residual tumor, a EQD2 of 70-77Gy is prescribed to GTV.
  Interventions: Radiation: RT

INTERVENTIONS:
Radiation: RT — All the patients receive extended resection to primary tumor and post-surgery RT. The patients are prescribed a EQD2 of 70-77Gy to GTV (residual tumor), 65-70Gy to CTV1(high-risk regions including tumor bed and gross macroscopic residual tumor), 50-55Gy to CTV2(low-risk regions) using Intensity-modulated radiotherapy (IMRT)

SUMMARY:
In China, mucosal melanoma of head and neck (MMHN) account for 30-40% of all melanoma and the incidence is on the rise. The prognosis of MMHN is poor with the 5-year survival in a range between 20-30%. The evidence for the treatment of MMHN was weak since large-sample clinical researches are rare and no prospective clinical trial is reported. Surgery is the primary treatment modality for MMHN. However, it is difficult to extend the necessary surgery range for MMHN due to its limitation of being adjacent to the important anatomical structure in head and neck or by the considerations of the protection for organ function. As a result, the recurrence rate for surgery along was over 50%. Radiotherapy(RT) is the main approach for the multidisciplinary treatment for MMHN. Benlyazid et al. conclude the data from 13 centers and find that compared to surgery alone, the addition of post-surgery RT improve the survival; The 5-year locoregional failure rate for the surgery alone group and the RT+surgery group were 55.6% and 29.9%, respectively. Currently, the research into the prognosis factors is spare for the non-metastatic MMMHN received extended resection to primary tumor. It is necessary to undertake a prospective clinical research for MMHN in the endemic area to estimate efficacy and safety of primary surgery plus postoperative radiotherapy with or without adjuvant chemotherapy, as well as to recognize the risk distribution in this cohort of patients, provide the evidence to improve the stratification treatment strategies in the clinic.

DETAILED DESCRIPTION:
All the patients enrolled are confirmed without any evidence of distant metastasis. All the patients receive extended resection to primary tumor and post-surgery RT. The patients are prescribed a EQD2 of 65-70Gy to CTV1 (high-risk regions including tumor bed), 50-55Gy to CTV2(low-risk regions) using Intensity-modulated radiotherapy (IMRT). The Prophylactic irradiation to upper neck is is decided by radiation physicians and given a EQD2 of 70-77Gy to CTVnd (clinically negative lymph nodes), 50-55Gy to CTVn2（neck nodal regions). If there is residual tumor, a EQD2 of 70-77Gy is prescribed to GTV. Adjuvant chemotherapy (for example, Temozolomide) is prescribed or not according the consideration of radiation physicians during RT or after RT. The clinical characteristics, radiation dose, chemotherapy regimen and the toxicities of are documented by the radiation physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed mucosal melanoma of head and neck (MMHN);
* Tumor staged as stages III/IVA (according to the American Joint Committee on Cancer 7th edition staging system) arising from head and neck according to the radiology and clinical exam;
* Prior local resection to primary tumor;
* Radiologically confirmed (MRI, CT or PET-CT if necessary) no regional lymph node present, nor any evidence of distant metastasis;
* Adequate marrow: white blood cell count of 4.0 × 109/L or more; absolute neutrophil of 2.0 × 109/L or more; haemoglobin concentrations of at least 90 g/L; platelet cell count of 100 × 109/L or more；
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 2.5×upper limit of normal (ULN)；
* Adequate renal function: creatinine clearance rate of more than 60 mL/min;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；
* Expected lifespan > 3 months;
* Patients must be informed of the investigational nature of this study and give written informed consent；
* Patients must be consent to the follow-up till death, the study termination or the end of the study.

Exclusion Criteria:

* Patients with histologically or radiologically distant metastasis or recurrence of primary tumor;
* Any contraception to RT;
* History of previous RT or chemotherapy;
* Any severe previous or intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, serious comorbidities, or had active lupus erythematosus or scleroderma, unstable cardiac disease needing treatment, chronic obstructive pulmonary disease exacerbation or other respiratory illness needing treatment, or an acute or fungal infection requiring treatmen);
* Prior malignancy within 5 years except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer;
* Pregnancy or lactation;
* Unable or unwilling to the compliance of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-07-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 3 year
  OS is calculated from the first day of therapy to the day of death, or to the last follow-up.

SECONDARY OUTCOMES:
Regional relapse-free survival(RRFS) | 3 Year
  RFS is calculated from the first day of therapy to regional failure from any cause. Regional relapses were diagnosed with clinical examination of the neck and, in doubtful cases, by fine needle aspiration or an MRI scan of the neck.
Local recurrence-free survival(LRFS) | 3 Year
  the first day of therapy to local failure from any cause. Local relapses were diagnosed by fibreoptic endoscopy and biopsy.
Distant metastasis-free survival (DMFS) | 3 Year
  DMFS is calculated from the first day of treatment to the date of first remote. Distant metastases were diagnosed by clinical symptoms, physical examinations, and imaging methods that included CT, MRI, bone scan, abdominal sonography, and/or PET-CT.
Number of participants with adverse events | 3 Year
  Number of participants with acute and late toxicity and treatment-related mortality.Adverse events were recorded according to the Common Terminology Criteria for Adverse Events (version 4.0) at each treatment visit, follow-up visit, and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: LiXia Lu, M.D., Study Chair — Sun Yat-sen University Cancer Center,China, Guangdong; LiXia Lu, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- LiXia Lu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandey M, Mathew A, Iype EM, Sebastian P, Abraham EK, Nair KM. Primary malignant mucosal melanoma of the head and neck region: pooled analysis of 60 published cases from India and review of literature. Eur J Cancer Prev. 2002 Feb;11(1):3-10. doi: 10.1097/00008469-200202000-00002. PMID 11917203
- [Background] Bishop KD, Olszewski AJ. Epidemiology and survival outcomes of ocular and mucosal melanomas: a population-based analysis. Int J Cancer. 2014 Jun 15;134(12):2961-71. doi: 10.1002/ijc.28625. Epub 2013 Dec 2. PMID 24272143
- [Background] McLaughlin CC, Wu XC, Jemal A, Martin HJ, Roche LM, Chen VW. Incidence of noncutaneous melanomas in the U.S. Cancer. 2005 Mar 1;103(5):1000-7. doi: 10.1002/cncr.20866. PMID 15651058
- [Background] Benlyazid A, Thariat J, Temam S, Malard O, Florescu C, Choussy O, Makeieff M, Poissonnet G, Penel N, Righini C, Toussaint B, Lacau St Guily J, Vergez S, Filleron T. Postoperative radiotherapy in head and neck mucosal melanoma: a GETTEC study. Arch Otolaryngol Head Neck Surg. 2010 Dec;136(12):1219-25. doi: 10.1001/archoto.2010.217. PMID 21173371
- [Background] Owens JM, Roberts DB, Myers JN. The role of postoperative adjuvant radiation therapy in the treatment of mucosal melanomas of the head and neck region. Arch Otolaryngol Head Neck Surg. 2003 Aug;129(8):864-8. doi: 10.1001/archotol.129.8.864. PMID 12925346
- [Background] Wu AJ, Gomez J, Zhung JE, Chan K, Gomez DR, Wolden SL, Zelefsky MJ, Wolchok JD, Carvajal RD, Chapman PB, Wong RJ, Shaha AR, Kraus DH, Shah JP, Lee NY. Radiotherapy after surgical resection for head and neck mucosal melanoma. Am J Clin Oncol. 2010 Jun;33(3):281-5. doi: 10.1097/COC.0b013e3181a879f5. PMID 19823070
- [Background] Bibault JE, Dewas S, Mirabel X, Mortier L, Penel N, Vanseymortier L, Lartigau E. Adjuvant radiation therapy in metastatic lymph nodes from melanoma. Radiat Oncol. 2011 Feb 6;6:12. doi: 10.1186/1748-717X-6-12. PMID 21294913
- [Background] Ballo MT, Garden AS, Myers JN, Lee JE, Diaz EM Jr, Sturgis EM, Morrison WH, Gershenwald JE, Ross MI, Weber RS, Ang KK. Melanoma metastatic to cervical lymph nodes: Can radiotherapy replace formal dissection after local excision of nodal disease? Head Neck. 2005 Aug;27(8):718-21. doi: 10.1002/hed.20233. PMID 15952196
- [Background] Morris KT, Marquez CM, Holland JM, Vetto JT. Prevention of local recurrence after surgical debulking of nodal and subcutaneous melanoma deposits by hypofractionated radiation. Ann Surg Oncol. 2000 Oct;7(9):680-4. doi: 10.1007/s10434-000-0680-y. PMID 11034246
- [Background] Frakes JM, Strom TJ, Naghavi AO, Trotti A, Rao NG, McCaffrey JC, Otto KJ, Padhya T, Caudell JJ. Outcomes of mucosal melanoma of the head and neck. J Med Imaging Radiat Oncol. 2016 Apr;60(2):268-73. doi: 10.1111/1754-9485.12404. Epub 2015 Nov 23. PMID 26597431
- [Background] Schild SE, Behl D, Markovic SN, Brown PD, Sande JR, Deming RL, Rowland KM Jr, Bearden JD. Brain metastases from melanoma: is there a role for concurrent temozolomide in addition to whole brain radiation therapy? Am J Clin Oncol. 2010 Dec;33(6):633-6. doi: 10.1097/COC.0b013e3181c4c54b. PMID 20042969
- [Background] Brachman DG, Pugh SL, Ashby LS, Thomas TA, Dunbar EM, Narayan S, Robins HI, Bovi JA, Rockhill JK, Won M, Curran WP. Phase 1/2 trials of Temozolomide, Motexafin Gadolinium, and 60-Gy fractionated radiation for newly diagnosed supratentorial glioblastoma multiforme: final results of RTOG 0513. Int J Radiat Oncol Biol Phys. 2015 Apr 1;91(5):961-7. doi: 10.1016/j.ijrobp.2014.12.050. PMID 25832688
- [Background] Middleton MR, Friedlander P, Hamid O, Daud A, Plummer R, Falotico N, Chyla B, Jiang F, McKeegan E, Mostafa NM, Zhu M, Qian J, McKee M, Luo Y, Giranda VL, McArthur GA. Randomized phase II study evaluating veliparib (ABT-888) with temozolomide in patients with metastatic melanoma. Ann Oncol. 2015 Oct;26(10):2173-9. doi: 10.1093/annonc/mdv308. Epub 2015 Jul 22. PMID 26202595
- [Background] Linardou H, Pentheroudakis G, Varthalitis I, Gogas H, Pectasides D, Makatsoris T, Fountzilas G, Bafaloukos D; Hellenic Cooperative Oncology Group. Predictive biomarkers to chemotherapy in patients with advanced melanoma receiving the combination of cisplatin--vinblastine--temozolomide (PVT) as first-line treatment: a study of the Hellenic Cooperative Oncology Group (HECOG). Anticancer Res. 2015 Feb;35(2):1105-13. PMID 25667500
- [Background] Guo J, Qin S, Liang J, Lin T, Si L, Chen X, Chi Z, Cui C, Du N, Fan Y, Gu K, Li F, Li J, Li Y, Liang H, Liu J, Lu M, Lu A, Nan K, Niu X, Pan H, Ren G, Ren X, Shu Y, Song X, Tao M, Wang B, Wei W, Wu D, Wu L, Wu A, Xu X, Zhang J, Zhang X, Zhang Y, Zhu H; written on behalf of Chinese Society of Clinical Oncology (CSCO) Melanoma Panel. Chinese Guidelines on the Diagnosis and Treatment of Melanoma (2015 Edition). Chin Clin Oncol. 2016 Aug;5(4):57. doi: 10.21037/cco.2015.12.02. Epub 2015 Dec 17. No abstract available. PMID 27164849
- [Background] Moreno MA, Roberts DB, Kupferman ME, DeMonte F, El-Naggar AK, Williams M, Rosenthal DS, Hanna EY. Mucosal melanoma of the nose and paranasal sinuses, a contemporary experience from the M. D. Anderson Cancer Center. Cancer. 2010 May 1;116(9):2215-23. doi: 10.1002/cncr.24976. PMID 20198705
- [Background] Burmeister BH, Mark Smithers B, Burmeister E, Baumann K, Davis S, Krawitz H, Johnson C, Spry N; Trans Tasman Radiation Oncology Group. A prospective phase II study of adjuvant postoperative radiation therapy following nodal surgery in malignant melanoma-Trans Tasman Radiation Oncology Group (TROG) Study 96.06. Radiother Oncol. 2006 Nov;81(2):136-42. doi: 10.1016/j.radonc.2006.10.001. Epub 2006 Oct 24. PMID 17064803
- [Background] Burmeister BH, Henderson MA, Ainslie J, Fisher R, Di Iulio J, Smithers BM, Hong A, Shannon K, Scolyer RA, Carruthers S, Coventry BJ, Babington S, Duprat J, Hoekstra HJ, Thompson JF. Adjuvant radiotherapy versus observation alone for patients at risk of lymph-node field relapse after therapeutic lymphadenectomy for melanoma: a randomised trial. Lancet Oncol. 2012 Jun;13(6):589-97. doi: 10.1016/S1470-2045(12)70138-9. Epub 2012 May 9. PMID 22575589
- [Background] Combs SE, Konkel S, Thilmann C, Debus J, Schulz-Ertner D. Local high-dose radiotherapy and sparing of normal tissue using intensity-modulated radiotherapy (IMRT) for mucosal melanoma of the nasal cavity and paranasal sinuses. Strahlenther Onkol. 2007 Feb;183(2):63-8. doi: 10.1007/s00066-007-1616-2. PMID 17294109
- [Background] Habermalz HJ, Fischer JJ. Radiation therapy of malignant melanoma: experience with high individual treatment doses. Cancer. 1976 Dec;38(6):2258-62. doi: 10.1002/1097-0142(197612)38:63.0.co;2-h. PMID 1000466
- [Background] Umeda M, Mishima Y, Teranobu O, Nakanishi K, Shimada K. Heterogeneity of primary malignant melanomas in oral mucosa: an analysis of 43 cases in Japan. Pathology. 1988 Jul;20(3):234-41. doi: 10.3109/00313028809059498. PMID 3060820
- [Background] Ballo MT, Ross MI, Cormier JN, Myers JN, Lee JE, Gershenwald JE, Hwu P, Zagars GK. Combined-modality therapy for patients with regional nodal metastases from melanoma. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):106-13. doi: 10.1016/j.ijrobp.2005.06.030. Epub 2005 Sep 22. PMID 16182463
- [Background] Poon I, Fischbein N, Lee N, Akazawa P, Xia P, Quivey J, Phillips T. A population-based atlas and clinical target volume for the head-and-neck lymph nodes. Int J Radiat Oncol Biol Phys. 2004 Aug 1;59(5):1301-11. doi: 10.1016/j.ijrobp.2004.01.038. PMID 15275713
- [Derived] Yao JJ, Zhang F, Zhang GS, Deng XW, Zhang WJ, Lawrence WR, Zou L, Zhang XS, Lu LX. Efficacy and safety of primary surgery with postoperative radiotherapy in head and neck mucosal melanoma: a single-arm Phase II study. Cancer Manag Res. 2018 Dec 14;10:6985-6996. doi: 10.2147/CMAR.S185017. eCollection 2018. PMID 30588103